CLINICAL TRIAL: NCT05257356
Title: Increased Emotional-motivational Processing in Patients with Chronic Pain and Its Neural Correlates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: susanne becker (Other)
Collaborators: SNSF (Unknown)
Responsible Party: Sponsor-Investigator, susanne becker, Head of Research Group, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: P000PS_203872/1
Record Dates: First submitted 2022-02-03; First posted 2022-02-25 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pain; Low Back Pain
Keywords: pain; chronic pain; emotional-motivational pain components; counterconditioning; negative hedonic shift
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Pain

STUDY DESIGN:
Intervention Model Description: Substudy 1(b): All participants will perform one psychophysical task to assess sensory-discriminative and emotional-motivational pain responses simultaneously. The responses and the reaction times of chronic pain patients will be compared to those of healthy participants to characterize possible alterations in the patients. Associative learning by monetary reinforcement will be implemented to diminish the aversiveness of the pain, which is assumed to be already increased in the patients.
  Substudy 2: As in Substudy 1, all participants will perform one psychophysical task to assess sensory-discriminative and emotional-motivational pain responses simultaneously combined with MRI assessing the effects of the counterconditioning on fronto-striatal circuits.
Who Masked: Participant
Masking Description: Participants are not fully instructed about the purpose before and during the test but will be debriefed after testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chronic Pain Patients (Experimental): All participants perform 1 psychophysical task to assess sensory-discriminative and emotional-motivational pain responses simultaneously. The performance of chronic pain patients will be compared to healthy volunteers to characterize possible alterations in patients. Associative learning by monetary reinforcement will be implemented to diminish the aversiveness of pain, which is assumed to be already increased in patients.
  Primary objectives: Show that emotional-motivational components are increased relative to sensory-discriminative components in chronic pain, and that enhanced emotional-motivational pain responses in chronic pain can be decreased by counterconditioning, leading to a normalization of pain perception relative to healthy individuals.
  Secondary objective: Assess whether chosen personality traits assessed by questionnaires can explain variations in sensory-discriminative and emotional-motivational pain responses.
  Interventions: Behavioral: psychophysical tasks
- Healthy Controls (Experimental): Substudy 1(b): Participants perform 1 psychophysical task to assess sensory-discriminative and emotional-motivational pain responses simultaneously. Associative learning by monetary reinforcement is implemented to diminish the pain aversiveness. Substudy2: Participants perform the same task combined with MRI assessing the counterconditioning effects on frontostriatal circuits.
  Primary objective: Show that emotional-motivational components are increased relative to sensory-discriminative components in chronic pain (Substudy 1(b)). Assess the neural correlates of the counterconditioning effects on emotional-motivational pain responses, specifically alterations in functional connectivity in frontostriatal networks compared to the unchanged natural state (Substudy 2).
  Secondary objective: To assess whether chosen personality traits assessed by questionnaires can explain variations in sensory-discriminative and emotional-motivational pain responses (Substudy1(b)+2).
  Interventions: Behavioral: psychophysical tasks

INTERVENTIONS:
Behavioral: psychophysical tasks — Substudy 1(b): All participants will perform one psychophysical task to assess sensory-discriminative and emotional-motivational pain responses simultaneously. The responses and the reaction times of chronic pain patients will be compared to those of healthy participants to characterize possible alterations in the patients (Substudy 1). Associative learning by monetary reinforcement will be implemented to diminish the aversiveness of the pain, which is assumed to be already increased in the patients.
  Substudy 2: As in Substudy 1, all participants will perform one psychophysical task to assess sensory-discriminative and emotional-motivational pain responses simultaneously combined with MRI assessing the effects of the counterconditioning on fronto-striatal circuits.

SUMMARY:
Chronic pain causes immense suffering and reductions in quality of life as well as enormous socioeconomic costs. Very many chronic pain patients fall into the category of unspecific pain, i.e. pain without clear medical explanation, with lacking effective treatments. It is assumed that a negative hedonic shift, characterized by excessive emotional-motivational processing and neg-ative affect, contributes causally to the development and maintenance of chronic pain. The mechanisms leading to such a shift are largely unclear; however, learning mechanisms appear likely candidates, possibly causing decreased connectivity in the fronto-striatal brain circuits. The project's over-all aim is to characterize mechanisms of emotional-motivational pain pro-cessing. The specific objectives are to illustrate that emotional-motivational pain components are heightened in chronic pain and that they can be de-creased by counterconditioning as an important and pervasive mechanisms in everyday life. Furthermore, its neural correlates in fronto-striatal networks underlying the conditioning effects will be characterized.

DETAILED DESCRIPTION:
Chronic pain is a major personal and societal problem causing immense suffering and reductions in quality of life as well as enormous socioeconomic costs (e.g. estimated as 11.2 Mio CHF of direct and indirect costs for chronic back pain in Switzerland in 2011. 90% of the chronic back pain patients fall into the category of unspecific pain, i.e. pain without clear medical explanation described as chronic primary pain in the new International Classification of Diseases ICD-11 (World Health Organization). This lack of medical explanation severely hampers diagnostic procedures and effective treatments. For such unspecific pain, strong influences of emotional and cognitive factors are known. However, the majority of pain research focuses on molecular and neuronal mechanisms of nociception (i.e. the neural encoding and processing of actually or potentially tissue-damaging events) without relating such processes to the subjective experience of and suffering from pain and modulatory psychological emotional-motivational influences. Considering the large category of unspecific pain and the fact that effective treatment is lacking, more research following a mechanism-oriented framework focusing on emotional-motivational pain components and related psychological mechanisms is needed, as done here.

The perception of pain is multidimensional: The International Association for the Study of Pain (IASP) defines pain as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage", highlighting the crucial point that pain always comprises emotional components. Specifically, pain comprises sensory-discriminative, emotional-motivational and cognitive-evaluative components as initially proposed in Melzack's tripartite model of pain. Typically, the sensory-discriminative and emotional-motivational components are well aligned; but these components can dissociate. For example, many people find a painful massage pleasant or enjoy eating hot chilies, likely through a reappraisal of the painful sensation. Extreme examples are prefrontal lobotomy, cingulotomy or strong morphine analgesia where pain is still recognized in its sensory-discriminative dimension, but loses its aversiveness and threat. Such a loss of emotional-motivational pain components can lead to severe injuries and life-threatening conditions. Although these examples affect only very few people, they illustrate a conceptually important point: Emotional-motivational aspects are the driving force in pain.

The dissociation of pain components: As described above and as an idea inherent to Melzack's tripartite model of pain, the different pain components can dissociate. The underlying mechanisms how such a dissociation can develop and be maintained are largely unclear. Based on earlier findings, operant and associative learning mechanisms appear to be likely candidates.

Applying the mechanisms of associative conditioning, a counterconditioning experiment showed impressively a dissociation between sensory-discriminative and emotional-motivational pain components. Counterconditioning is a specific form of classical conditioning used to reduce negative stimulus valence through a new association between a behavior and a stimulus of an oppositive valence. For example, Eroféeva applied this principle in the context of pain, pairing a positive stimulus (food) with an aversive painful stimulus in dogs. The appetitive response to the positive stimulus gradually and completely replaced aversive pain responses, suggesting that the pain lost its aversiveness, thus diminishing its emotional-motivational component. However, since the dogs still utilized the painful stimulus to predict the rewarding stimulus, sensory-discriminative pain components must have been preserved. This example illustrates that learning might be a mechanism underlying a gradual dissociation of sensory-discriminative and emotional-motivational pain components.

The negative hedonic shift in chronic pain: In line with the observation that learning related to a dissociation of different pain components can be altered, emotional-motivational components appear to dominate over sensory-discriminative components in chronic pain. For example, the influential Fear-Avoid-ance Model of Pain termed chronic pain as "exaggerated pain perception" in its earliest version, because of disproportionally augmented emotional-motivational relative to sensory-discriminative pain components. Such increased emotional-motivational pain perception is often reflected in chronic pain patients in heightened pain aversiveness and pain avoidance behavior. Further and in line with such increases, recent findings suggest that pain processing is characterized by a functional shift from nociceptive to non-nociceptive emotional brain circuits in chronic pain, specifically to fronto-striatal circuits. Such a shift in chronic pain fits the observation of augmented negative affect and impaired motivated behavior, mirrored in anhedonia (i.e. the inability to feel pleasure) and very high comorbidity (up to 86%) between chronic pain and affective disturbances. Based on such observations, chronic pain has been described to induce a negative hedonic shift. Although this suggestion has been cited often and is compelling in explaining the development and maintenance of unspecific chronic pain, the underlying mechanisms of such a shift have not directly been investigated so far. It has been shown that patients with constant chronic back pain have increased activation in the medial prefrontal cortex (mPFC) and in the amygdala, as well as an increased incidence of white matter and increased functional connections between the mPFC, the nucleus accumbens (NAcc) and the amygdala compared to recovered patients and healthy controls. Of particular importance, altered fronto-striatal circuits, especially the increased functional connectivity between the NAcc and ventromedial prefrontal cortex (vmPFC), predicts the transition from subacute to chronic pain. Moreover, the importance of the NAcc-vmPFC connectivity for the modulation of pain perception has been confirmed in healthy persons.

The aims of this study are therefore (1) to illustrate that emotional-motivational components are in-creased relative to sensory-discriminative components in chronic pain, (2) to show that increased emo-tional motivational pain responses in chronic pain can also be decreased by counterconditioning, leading to a normalization of pain perception relative to healthy individuals as well, and (3) to assess the neural correlate of the counterconditioning effects on emotional-motivational pain responses, specifically alterations in functional connectivity yin fronto-striatal networks.

Intended intervention: All participants perform one psychophysical task to assess sensory-discriminative and emotional-motivational pain responses simultaneously. In Substudy 1 an associative learning paradigm will be implemented to dissociating the sensory-discriminative pain responses compared to emotional-motivational pain responses by monetary reinforcement. In Substudy 2, the effects of the counterconditioning on fronto-striatal networks will be assessed by MRI.

Potential for new scientific generalizable knowledge: Our knowledge on the basic mechanisms of pain increased rapidly in recent years. Nevertheless, treatment of chronic pain is surprisingly unsuc-cessful. Particularly, patients suffering from unspecific pain often do not get efficient treatment. This gap between basic knowledge and applied treatment likely is caused by a mismatch between research foci and the subjective complains of patients. Basic research focuses on neurobiological basic mechanisms, e.g. on molecular and neuronal levels. Although indisputable of high relevance for our understanding of pian, it is hard to transfer these basic mechanisms directly to the multifaceted experience of pain in humans, because this can be strongly modulated by emotional and cognitive processes. The goal of this study is to provide a substantial contribution to lose this gap by (1) providing new methods needed for an appropriate investigation of the problem outlined and (2) by gathering new knowledge on pain mechanisms relevant in the development and maintenance of chronic pain.

This study is a Clinical Study Category A because it includes an intervention that is neither a drug nor a transplant. The risk for the participants is minimal.

ELIGIBILITY:
HEALTHY PARTICIPANTS

Inclusion criteria:

* Between 18 and 70 years of age (in Substudy 1: age- and sex-matched to chronic pain patients)
* Good overall health status
* Sufficient knowledge of German or English to follow instructions
* Ability to give written informed consent

Exclusion criteria:

* Pain longer than >3 consecutive days and on more than 30 days within the last 12 months
* Major psychiatric or neurological disorders, and substance abuse
* Consumption of alcohol, illegal drugs, and analgesic drugs within 24 hours before testing
* Pregnancy
* For Substudy 2: An MR-specific safety questionnaire will be filled in to check for any contradiction to magnetic resonance imaging (MRI): wearing an electronic device, implants or prosthetics, injury from metal parts or fragments, metal parts in or on the body, surgery on the head, heart or back, tattoo or permanent makeup, problems lying still for long periods of time, claustrophobia, possible pregnancy, metal contraceptive coil

CHRONIC PAIN PATIENTS

Inclusion criteria:

* Between 18 and 70 years of age
* Unspecific musculoskeletal pain as defined according to the ICD-11 as chronic primary pain (MG30.1, e.g. chronic widespread pain, complex regional pain syndrome, chronic primary headache or orofacial pain, chronic migraine, chronic tension-type headache, trigeminal autonomic cephalalgias, burning mouth syndrome, chronic primary visceral pain, irritable bowel syndrome, chronic primary musculoskeletal pain), and which is not classified as chronic cancer related pain (MG30.2; e.g. chronic cancer pain, chronic post-cancer treatment pain), chronic postsurgical or post traumatic pain (MG30.3; e.g. chronic postsurgical pain, chronic posttraumatic pain), chronic secondary musculoskeletal pain (MG30.4; e.g. chronic musculoskeletal pain from persistent inflammation, chronic musculoskeletal pain associated with structural changes, chronic musculoskeletal pain associated with a disease of the nervous system), chronic secondary visceral pain (MG30.5; e.g. chronic visceral pain from persistent inflammation, chronic visceral pain from vascular mechanisms, chronic visceral pain from mechanical factors), chronic neuropathic pain (MG30.6; e.g. chronic peripheral neuropathic pain, trigeminal neuralgia, postherpetic neuralgia, chronic central neuropathic pain), chronic secondary headache or orofacial pain (MG30.7; e.g. chronic dental pain, chronic neuropathic orofacial pain, trigeminal neuralgia, headache or orofacial pain attributed to chronic secondary temporo-mandibular disorders), other specified chronic pain (MG30.Y), or other non-specified chronic pain (MG30.Z)
* Sufficient knowledge of German or English to follow instructions
* Ability to give written informed consent

Exclusion criteria:

* Major psychiatric or neurological disorders, and substance abuse
* Regular intake of opioids for pain (e.g. burprenorphine, codeine, fentanyl, hydromorphone, orphine, oxycodone, tapentadol, tilidine/na-loxone, tramadol)
* Consumption of alcohol, illegal drugs, and analgesic drugs within 24 hours before testing
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Successful Avoidance Responses | during the procedure
  In Substudy1(b) and Substudy2: The number of successful avoidance responses upon correct discrimination responses in the task assessing sensory-discriminative and emotional-motivational pain responses simultaneously.
Fronto-striatal Networks | during the procedure
  In Substudy 2: Blood oxygen level dependent (BOLD) signal and changes in functional connectivity in fronto-striatal networks while assessing sesnorydiscriminative and emotional-motivational pain responses simultaneously.

SECONDARY OUTCOMES:
Reaction Times (RT) | during the procedure
  reaction times (RT) in the trials of the psychophysical task
Pain Threshold in °C | baseline
  individual pain threshold assessed with experimental heat pain by the methods of limits
Pain Tolerance in °C | baseline
  individual pain tolerance assessed with experimental heat pain by the methods of limits
Visual Analogue Scale (VAS) for Perceived Pain Intensity | during the procedure
  self-reported perceived pain intensity assessed with experimental heat pain rated on a visual analogue scale (VAS) from 0 (no sensation) to 100 (pain threshold) and 200 (most intense pain tolerable)
Visual Analogue Scale (VAS) for Perceived Pain Unpleasantness | during the procedure
  self-reported perceived pain unpleasantness assessed with experimental heat pain rated on a visual analogue scale from -100 (extremely unpleasant) to 0 (neutral) and +100 (extremely pleasant).
Fear of Pain Questionnaire (FPQ-III) Score | during the procedure
  assessing pain-related fear; rating 30 items on a five-point Likert scale from 1 = "not afraid at all" to 5 = "extremely afraid"
Fear-Avoidance Beliefs Questionnaire (FABQ) Score | during the procedure
  assessing fear of pain and the resulting avoidance of physical activity or work; rating 16 items on a seven-point Likert scale from 0 = "completely disagree" to 5 = "completely agree"
Pain Catastrophizing Scale (PCS) Score | during the procedure
  assessing thoughts and feelings when experiencing pain (catastrophizing); rating 13 items on a five-point Likert scale from 0 = "not at all" to 4 = "all the time"
Need Inventory of Sensation Seeking (NISS) Score | during the procedure
  assessing sensation seeking as a motivational trait; rating 17 items on a five-point Likert scale from 1 = "almost never" to 5 = "almost always"
Revised Life-Orientation Test (LOT-R) Score | during the procedure
  assessing dispositional optimism; rating 10 items on a five-point Likert scale from 0 = "strongly disagree" to 4 = "strongly agree"
Snaith-Hamilton Pleasure Scale (SHAPS) Score | during the procedure
  assessing individual hedonic capacity; rating 14 items with a set of 4 response categories "definitely agree", "agree", "disagree" and "strongly disagree", with either of the agree responses receiving a score of 0, and with either of the disagree responses receiving a score of 1
Short Form of the Barratt Impulsiveness Scale (BIS-15) Score | during the procedure
  assessing the personality trait of impulsivity; rating 5 items on a four-point Likert scale from 1 = "rarely / never" to 5 = "almost always / always"
West Haven-Yale Multidimensional Pain Inventory (WHYMPI) Score | during the procedure
  assessing clinical pain and pain chronicity; rating 20 items with a set of 7 response categories (scores from 0 to 6), with higher values indicating higher clinical pain and pain chronicity
Autonomic Reactions: Electrocardiography (ECG) | during the procedure
  assessing changes in the heart rate via electrocardiography (ECG) as an indicator of sympathetic activities in response to the pain stimuli and task performance
Autonomic Reactions: Galvanic Skin Response (GSR) | during the procedure
  assessing changes in the skin conductance with via Galvanic Skin Response (GSR) as an indicator of sympathetic activities in response to the pain stimuli and task performance

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Becker, Dr. Prof., Principal Investigator — Balgrist Universitätsklinik
Locations (1):
- Balgrist Campus, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No